CLINICAL TRIAL: NCT01854294
Title: GM604 Phase 2A Randomized Double-blind Placebo Controlled Pilot Trial in Amyotrophic Lateral Disease (ALS)
Acronym: GALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genervon Biopharmaceuticals, LLC (Industry)
Collaborators: Columbia University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GALS 001
Record Dates: First submitted 2013-05-08; First posted 2013-05-15 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2019-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; motorneuron disease; Central Nervous System (CNS) disease; neurodegeneration; neuroprotective; mechanisms of action; pathways; biomarkers; Cerebral Spinal Fluid (CSF); blood biomarkers; multi-factorial; multisystem; single target; pathogenic mechanisms; Protein Bands Selection by Function; in silico analysis; active site; protein; peptide; embryonic stage; endogenous; master regulators; fetal development; embryonic development; common pathways; Blood Brain Barrier (BBB); anti-inflammatory; anti-apoptotic; anti-oxidative; regenerative; distress signals; neurotrophin; Motoneuronotrophic factor (MNTF); ALS model; life span; disease onset; grip strength; protein expression; DNA microarray; differential expression; Phase 1 clinical trial; rare disease; common underlying pathogenic mechanisms; neurological deficits; gene mutation; misfolded proteins; inadvertent errors; modulation of genes; master regulator peptide drug; ALS related genes; mitochondria dysfunction; excitotoxicity; axonal transport; oxidative stress; protein aggregation; pathogenesis; target biomarkers; efficacy biomarkers
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Central Nervous System Diseases; Nerve Degeneration; Rare Diseases; Mitochondrial Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GM604 treated (Experimental): 8 subjects will receive GM604. Each GM604 treated subject will receive a slow IV bolus injection (~1min) of 6.4 mL (320mg @50 mg/mL=6.4 mL) for each dose. A total of 6 doses will be administered over two weeks (on Mondays, Wednesdays and Fridays for the first 2 weeks).
  Interventions: Drug: GM604
- Placebo comparator (Placebo Comparator): 4 subjects will receive placebo. 6.4 mL Bacteriostatic saline will be used for the Placebo group. Injections will be given to the subject in the same manner as in GM604 treated group. A total of 6 doses will be administered over two weeks (on Mondays, Wednesdays and Fridays for the first 2 weeks).
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: GM604 — GM604 treated group subject will receive a slow IV bolus injection (~1min) of 6.4 mL (320mg @50 mg/mL=6.4 mL) for each dose. A total of 6 doses will be administered over two weeks (on Mondays, Wednesdays and Fridays for the first 2 weeks).
  Other Names: GM6; GM602; GM608
  Arms: GM604 treated
Drug: Placebo comparator — Placebo comparator group subject will receive a slow IV bolus injection (~1min) of 6.4 mL bacteriostatic saline for each dose. A total of 6 doses will be administered over two weeks (on Mondays, Wednesdays and Fridays for the first 2 weeks).
  Other Names: Bacteriostatic saline
  Arms: Placebo comparator

SUMMARY:
GM604 is an endogenous human embryonic stage neural regulatory and signaling peptide that controls the development, monitoring and correction of the human nervous system. Neurological diseases are multisystem, multifactorial, and single target drugs are ineffective. Genervon's Master Regulators play a significant role in embryonic/fetal nervous system development and are potent disease modification drug candidates modulating many pathways including inflammation, apoptotic, and hypoxia. The study drug is an regulatory peptide with a sequence identical to one of the active sites of human Motoneuronotrophic Factor and is manufactured by solid phase synthesis. Pre-clinical research indicates it to be a neuro-protective agent in animal models of ALS, motorneuron diseases, PD, other neuro-degenerative diseases and stroke. GM604 controls and modulates over many known and significant ALS genes with positive effects interactively and dynamically through multiple pathways, and up to twenty-two biological processes, including neuro-protection, neurogenesis, neural development, neuronal signaling, neural transport, and other processes. GM6 is not a cocktail of drugs, but one master regulator peptide drug that functions through multiple pathways. Genervon hypothesized that studying the biomarkers of protein expressions of these ALS genes such as superoxide dismutase 1 (SOD1) and the protein expression of substances such as tau, neurofilament - heavy (NF-H), Cystatin C which were indications of degeneration of neuron in the CSF collected from ALS patients will provide information of the possible GM604's mechanisms of action in treating ALS. 1. This pilot trial is designed to test proof of principle, i.e. determine if a 2-week IV bolus treatment with this agent can (1) change ALS protein expression (target biomarkers and efficacy biomarkers) after treatment (2) have preliminary effects measures of ALS disease clinical progression.

Study Objectives are:

1. To test the safety and tolerability of GM604 in a population of ALS patients.
2. To test for changes in ALS biomarkers before and after treatment.
3. To determine preliminary effects of injections of GM604 on measures of ALS disease biomarkers and clinical progression

DETAILED DESCRIPTION:
Background

1. In the early 1990s Genervon hypothesized that Central Nervous System / Peripheral Nervous systme (CNS/PNS) and rare motoneuron diseases and disorders involve the interplay of a highly complex, multifactorial process of many non-dominant effectors in an interactive dynamic network. Therefore Genervon decided for its drug development strategy the classic single target drug development paradigm is not likely leading to a cure.
2. Genervon also hypothesized that aging is likely the initial multifactorial triggers that lead to multiple defective or degraded gene products accumulating with advancing years. However the key to a cure for many human neurological disorders is in the subsequent common terminal cascade coinciding with the onset of neurological deficits. The terminal cascade involves the shared pathways of interactive multifactorial pathogenic mechanisms that lead to the ultimate demise of neurons. Therefore Genervon's strategy is not to find the triggers or the residue debris of neuron death in discrete areas of the central nervous system.
3. Genervon recognized the limited human capacity to design a drug that can dynamically and interactively modulate multiple pathways and genes. Therefore one possible drug development strategy is to find the endogenous early stage regulatory molecule(s) that controls the development, monitoring and correction of the human nervous system.
4. Genervon developed a novel proprietary technology platform named Protein Bands Selection by Function to find the fetal signal regulators. One of the discoveries is a 33 amino acid peptide we named human Motoneuronotrophic Factor (MNTF), its gene sequence and its chromosome location.
5. Genervon developed another novel platform named In Silico Analysis to find active sites within bigger proteins. Within the MNTF peptide, Genervon identified a family of nine embryonic stage human multifactorial master regulators which govern nervous system development, protection and correction. These master regulators are highly expressed in week 9 of embryonic/fetal development, a time of incredible intricacies, but truly remarkable consistency as well.
6. Genervon has developed one of the nine master regulators named GM6 for disease modification of CNS/PNS and neurodegenerative diseases and disorders with shared or common pathways of interactive multifactorial pathogenic mechanisms. GM6 binds to Insulin Receptor beta sub-unit and Insulin Growth Factor Receptor 1 and Receptor 2 (IGF1R/IGF2R) which also have the identical sub-unit. GM6 penetrates the Blood Brain Barrier (BBB) and activates many appropriate genes through multiple pathways to induce anti-inflammatory, anti-apoptotic, anti-oxidative and regenerative effects in response to the dynamic distress signals from the nervous system.
7. GM6 is also known as GM604, GM602 and GM608. Drug name GM604 is assigned to ALS indication. GM602 is assigned to stroke indication. GM608 is assigned to Parkinson Disease indication.
8. The investigational drug GM604 is a regulatory/signaling peptide with a sequence identical to one of the nine active sites of human Motoneuronotrophic factor (MNTF), also referred to as GM6 in studies. MNTF is a novel human endogenous developmental stage neurotrophin for the nervous system with a specific human chromosome location.
9. Pre-clinical efficacy studies: The investigators' preclinical animal study has shown that intravenously injected GM604 is able to penetrate the blood-brain barrier and enter the brain. GM604 has shown neuroprotection in a variety of in vitro and animal models of numerous CNS diseases including ALS, ischemic stroke, spinal cord injuries, Parkinson's disease (PD), multiple sclerosis (MS), Alzheimer Disease (AD) and Huntington Disease (HD).
10. GM6 provided neuroprotection for neurons in vitro against soluble inflammatory factors in human CSF from patients with various CNS diseases. It increased neurons survival by 175% after exposure to ALS patients' CSF, by 191% in AD patients' CSF, by 198% in PD patients' CSF, by 205% in Stroke patients' CSF, by 246% in MS patients' CSF and by 273% in HD patients' CSF.
11. Preclinical research in animal models indicates GM604 to be a neuroprotective agent in animal models of ALS, motoneuron disease, Parkinson's disease and stroke. In ALS model, SOD1 mice from Jackson Lab stock #G93A were treated with GM604 at 0, 1 and 5 mg/kg. SOD1 mice were examined for age of disease onset, age of death, and behavioral expression of the disease (CS=Clinical score). GM604 prolonged life span in ALS mice SOD1 by 30% [(163.5-126)/126 = 30%], delayed median clinical score by 53%, delayed symptoms onset by 27% [(145.5-114.5)/114.5 = 27%] at 5 mg/kg dose. The conclusion is that GM6 significantly showed a dose dependent effect in delaying age of onset of the disease, age of death, increasing grip strength and rota-rod performance, and improving clinical score of the treated animals.
12. The investigators found out later in the study of Wobbler Mouse model that the optimal dose for SOD1 mice model should probably be 20 mg/kg and will probably see even more significant effects if 20 mg/kg were used in the SOD1 mice study.
13. GM604 20mg/kg dramatically increased the survival life span by 500% (6 fold from 7-14 weeks to 55-65 weeks) and the control animals and animals treated with low doses of GM6 showed a continual decrease in grip strength. Wobbler mice treated with GM6 at 10-20 mg/kg showed an improvement in grip strength out to 4 weeks (3 fold). GM604 10 and 20 mg/kg treatment showed a significant increase in body weight out to 8 weeks following treatment.GM604 10 and 20 mg/kg treatment increased of preservation of motor neurons by 160% (2.6 fold).

The conclusion is that GM604 was found to be efficacious in an in vivo mouse model of neurological disease. The effectiveness of GM604 was dose-dependent and indicates that GM604 may be beneficial in treating various neurological disorders.

Rationales

1. This pilot trial is designed to test proof of principle, i.e. determine if a 2-week IV bolus treatment with this agent can (1) change ALS protein expression (target biomarkers and efficacy biomarkers) after treatment (2) have preliminary effects measures of ALS disease clinical progression.
2. Previous human experience: A Phase 1 Clinical Trial Study has been completed. The Phase 1 Trial primary objective is to determine the safety and tolerability and to establish the pharmacokinetic and pharmacodynamic properties of GM602 at 0.5, 1.5, and 5.0 mg/kg administered as a single bolus intravenous dose in human subjects and after 3 consecutive daily doses of GM602 at the highest safe and tolerated dose of 5.0 mg/kg. The Phase 1 study established that 3 consecutive daily doses of 5.0 mg/kg of GM602 are safe and tolerated.
3. Concurrently, other Investigational New Drug (IND) and on-going clinical trials with GM6 are:

IND 77,789: "A Phase 2 double blinded, randomized, placebo controlled dose escalation Study to Evaluate the Efficacy and the Safety of GM602 in Patients with Acute Middle Cerebral Artery Ischemic Stroke within an 18 h-hour treatment window. Acronym/Title is GMAIS. GM602 received fast track designation for ischemic stroke in 2007. The stroke trial has not completed enrollment and has not unblinded the treatment randomization to generate drug related safety report.

IND 109,441: "GM602 in A Phase IIA Pilot double-blinded, randomized, placebo controlled trial in mild to moderate Parkinson Disease (PD). Acronym/Title is GAP-PD. The PD trial is recruiting patients.

Possible GM604 Mechanisms of Action (MOA) in ALS

1. More and more scientists are publishing papers advocating that ALS is a multifactorial disease. Other rare diseases including CNS/PNS diseases and disorders are multifactorial and multisystem diseases as well, i.e. multiple interactive biologic systems and genes are compromised and failing like domino.
2. One of the major reasons for CNS clinical trials that have uniformly failed is that the classic drug development paradigm of designing single target drug for CNS/PNS and rare diseases' pathogenesis simply would not be able to handle the multifactorial nature of the complex diseases.
3. An initial trigger(s) which is likely to be multifactorial and cumulative is followed by a terminal cascade which also involves interactive multifactorial pathogenic mechanisms, coinciding with the onset of neurological deficits, genes mutation and or expression of misfolded proteins. That is simply why a single target drug is not able to do the job. Most neurological diseases and disorders have common underlying pathogenic mechanisms that lead to neural death. Our drug development strategy is to find an endogenous regulator to interactively and dynamically modulate these common underlying pathogenic mechanisms.
4. Genervon changed the drug development paradigm from hitting a single gene/pathway to a comprehensive and dynamic, multifactorial approach to treat complex rare and neurodegenerative diseases with a multi-factorial drug GM604. GM604 is one of the embryonic/fetal stage MNTF master regulators that is an endogenous signaling peptide for the development and regulations of the nervous system development. GM604 is multifactorial and corrects inadvertent errors in embryonic/fetal development and this neuroprotection and correction property may be applied to neurodegenerative disease therapy in adults.
5. Genervon studied the mechanisms of action of GM6 by DNA microarray technique. GM604 controls and modulates many known and significant ALS genes with positive effects, through multiple pathways interactively, systemically and dynamically. Our master regulator peptide drug modulates not just one but many ALS related genes. It is not a cocktail of drugs, but one master regulator peptide drug.
6. Mechanisms that have been postulated in ALS are a complex interplay between multiple pathogenic processes including oxidative stress, protein aggregation, mitochondrial dysfunction excitotoxicity, and impaired axonal transport. GM604 modulates genes involved in these pathways and others. Genervon has also identified some genes to be tested as targets.
7. ALS is notoriously fatal and has many alternate forms with different pathogenesis. Therefore all the previous single target drug trials have to restrict the enrollment to very small selective segment of ALS patients. With the potential that GM604 functions through multiple pathways and modulate multiple ALS related genes, Genervon believes GM604 can potentially treat ALS patients from a variety of segments instead of restricting to small selective segment of ALS patients. Genervon is proposing an ALS Phase 2 clinical trial that is broadly inclusive.

Use of Biomarkers for ALS

Most late-phase clinical trials across all diseases fail to demonstrate drug efficacy between case and controls. The incorporation of biomarkers within clinical trials may reduce this 'drug attrition' rate. The biomarkers to be incorporated into clinical trials can be subdivided into:

1. 'Target' biomarkers (the drug hits its target and, therefore, provide benefit),
2. 'Efficacy' biomarkers (indicators of positive drug effect (result) via the mechanism of drug action).
3. 'Efficacy/Target biomarkers.

Genervon hypothesized that modulating disease causing genes may modulate ALS disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ALS: Familial and Sporadic ALS, with symptom onset < or equal to 24 months.
2. At least 18 years of age
3. Subjects meet the El Escorial criteria of definite criteria for a diagnosis of ALS.
4. Subjects can be on a stable dose of riluzole for at least a month or not taking or initiating riluzole for the duration of the trial.
5. Not on any experimental medication for the last 1 month or five times the half-life of experimental medication.
6. At screening, must have a Forced Vital Capacity (FVC) ≥ 65% of predicted capacity for age, height and gender.
7. Have fully completed informed consent form
8. Ability to comply with study procedures
9. Women of child-bearing age must be on birth control. Pregnancy test should be done in women in child bearing age.
10. Medically safe to have lumbar puncture to collect CSF

Exclusion Criteria:

1. History of liver disease, severe renal failure, diabetes, coronary heart disease, cancer
2. Clinically significant EKG abnormality at screening
3. Any comorbid condition which would make completion of the trial unlikely
4. FVC < 65%
5. Presence of a bleeding disorder
6. Allergy to local anesthetics
7. Problem with CSF pressure
8. Topical or other skin infection at the lumbar puncture site
9. BMI > 32 kg/m2
10. Medical or surgical conditions in which a lumbar puncture is contraindicated
11. Use of any anti-platelet or anticoagulant drugs, such as plavix, aggrenox, ticlid, warfarin or coumadin

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Efficacy by percent change in biomarker in th CSF at week 12 from baseline | baseline, week 2, week 12
  Efficacy by percent change in biomarker in the CSF at week 12 from baseline: (a) Efficacy biomarkers (b) Target biomarkers (c) Efficacy/target biomarkers
Safety by measuring 1. adverse event frequency and severity, changes in vital signs, clinical laboratory values. 2. Serious adverse event frequency | baseline, week 2, week 12
  Safety: 1. adverse event frequency and severity, changes in vital signs, clinical laboratory values. 2. Serious adverse event frequency
Tolerability by measuring the ability to complete the first 2 weeks of active treatment in the study | Baseline, week 2, week 12
  Tolerability: The ability to complete the first 2 weeks of active treatment in the study

SECONDARY OUTCOMES:
ALSFRS-R (Amyotrophic Laeral Sclerosis Functional Rating Scale - Revised) | Symptom onset, screening, baseline, week 2, week 6, week 12
  Progressive change in ALSFRS-R of each patient determined from the following data points:1) symptom onset, 2) baseline, 3) end of week 2 examination, 4) end of week 6 examination and 5) end of week 12 examination.
Forced Vital Capacity (FVC) | Symptom onset, baseline, week 2, week 6, week 12
  Progressive change in Forced Vital Capacity (FVC) from the following data points: 1) symptom onset, 2) baseline, 3) end of week 2 examination, 4) end of week 6 examination and 5) end of week 12 examination.
Time Up and Go (TUG) | Symptom onset, baseline, week 2, week 6, week 12
  Progressive change in Forced Vital Capacity (FVC) from the following data points: 1) symptom onset, 2) baseline, 3) end of week 2 examination, 4) end of week 6 examination and 5) end of week 12 examination.
muscle strength | Symptom onset, baseline, week 2, week 6, week 12
  Progressive muscle strength change measured by HHD (handheld dynamometry testing score) from the following data points: 1) symptom onset, 2) baseline, 3) end of week 2 examination, 4) end of week 6 examination and 5) end of week 12 examination.
Biomarker in blood | baseline, week 2, week 6, week 12
  Percentage changes in Biomarkers in blood between baseline and 1) the end of week 1, 2) end of week 2, 3) end of week 6 and 4) end of week 12. Comparing the changes encompassing the entire cohort of 10 subjects.
Mortality rate | baseline, week 2, week 6, week 12
  Report all death as mortality rate

OTHER OUTCOMES:
comparison of slopes (change in the rate of decline)of disease progression | Symptom onset, baseline, week 2, week 6, week 12
  Secondary analyses may consider a comparison of slopes (change in the rate of decline) for any hint of disease modification using placebo outcomes in patients matched for baseline features from a large database of recent clinical trials by NEALS showing stable rates of decline as historical controls.
stratification of patients by symptoms | Symptom onset, baseline, week 2, week 6, week 12
  Secondary analysis to allow a-priori stratification of patients by their symptoms if available
  1. predominantly lower motor neuron
  2. predominantly upper motor neuron
  3. predominantly bulbar

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Mitsumoto, MD, Principal Investigator — Columbia Medical Center NY; Merit Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia Medical Center NY, New York, New York